CLINICAL TRIAL: NCT04434209
Title: Limiting AKI Progression in Sepsis (LAPIS): a Phase 4, Multicenter, Randomized Controlled Trial of Biomarker-guided Delivery of Kidney-sparing Care Measures in Sepsis Subjects At Risk of Developing AKI
Brief Title: A Study Looking At the Use of Biomarkers to Provide Early Indication of Acute Kidney Injury in Patients with Sepsis (Limiting AKI Progression in Sepsis)
Acronym: LAPIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Highly improbable to reach recruitment objective due to impact of COVID-19 pandemic
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LAPIS
Record Dates: First submitted 2020-05-26; First posted 2020-06-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Acute Kidney Injury; Septic Shock
Keywords: Sepsis; Acute Kidney Injury; Kidney damage; Septic shock; Biomarkers
MeSH Terms: conditions — Sepsis; Acute Kidney Injury; Shock, Septic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NephroCheck-guided interventions (Experimental)
  Interventions: Device: Subject management guided by NephroCheck® test
- Standard of Care (Active Comparator): Standard of Care assessment and treatment
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Subject management guided by NephroCheck® test — NephroCheck® is a device using biomarkers to identify subjects at risk of sepsis-associated acute kidney injury
  Arms: NephroCheck-guided interventions
Other: Standard of Care — Standard of Care patient management
  Arms: Standard of Care

SUMMARY:
Biomarkers that provide an early indicator of kidney stress could be useful in clinical practice to detect silent episodes of acute kidney injury (AKI) or for early identification of subjects at risk of AKI. Two urinary biomarkers have been identified as early indicators of AKI. The NephroCheck® test is a commercially available test that uses these biomarkers, and this study assesses the use of these in reducing negative clinical outcomes for patients with sepsis-associated AKI. The study will enroll subjects diagnosed with sepsis, including septic shock, who will be randomly assigned to either receive NephroCheck®-guided kidney-sparing and fast-tracking interventions; or to receive current Standard of Care assessment and treatment.

NOTE: Participants are no longer being recruited to this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sepsis or septic shock.
* Admission to the ICU or planned admission to the ICU with an expected stay of 72 hours or more after enrollment in the same hospital.
* Expected to have indwelling urinary catheter placed and kept until at least 48 hours after enrollment.
* Written informed consent.

Exclusion Criteria:

* Women with known pregnancy, prisoners or institutionalized individuals.
* Previous renal transplant.
* Stage 2 or 3 Acute Kidney Injury (AKI) at screening.
* Receiving dialysis (either acute or chronic), or in imminent need of dialysis at enrollment.
* Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2.
* Known End Stage Renal Disease (ESRD) or history of active nephrotic syndrome within the last 3 months.
* Known Stage 2-3 AKI within last 2 weeks.
* Terminally ill (defined as expectation of death within 6 months), has a do not resuscitate order that would restrict protocol-required procedures, or is being admitted only for palliative care.
* History of solid organ transplant and receiving calcineurin inhibitors.
* Documented serious allergy (i.e. anaphylaxis) to vancomycin, aminoglycosides, penicillins, or cephalosporins (intravenous or oral).
* Known current serum total bilirubin > 4mg/dL.
* Subjects already included in an observational study can be co-enrolled in LAPIS. Subjects already included in an interventional study may be enrolled with pre-approval of the sponsor according to the following rules:

  1. Co-enrollment in LAPIS will not be allowed with investigational drug and device studies;
  2. Studies may be allowed if AKI or kidney function is not an endpoint with pre-approval of the LAPIS sponsor;
  3. Co-enrollment in LAPIS will not be allowed if co-enrollment is an exclusion criterion in the other study.
* Subjects with laboratory confirmed COVID-19 infection as the primary reason for hospital admission.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Number of deaths, dialysis or progression of AKI | Enrollment to 72 hours
  Measured by composite number of deaths, dialysis or progression of AKI. Dialysis defined as any form of renal replacement therapy (RRT); progression of AKI defined as Stage 0 to 2/3 or Stage 1 to 3.

SECONDARY OUTCOMES:
Number of participants with progression of AKI | Enrollment to 48 and 72 hours
  Progression of AKI (Acute Kidney Injury) to Stage 2 or 3 during the time frame. Measured independently.
Number of deaths | Enrollment to 48 and 72 hours
  Number of deaths. Measured independently.
Number of participants receiving dialysis | Enrollment to 48 and 72 hours
  Dialysis defined as any form of renal replacement therapy (RRT). Measured independently.
Number participants at Stage 2 or 3 AKI | Enrollment to 72 hours
  Defined as highest stage of AKI during the time frame
ICU length of stay | Enrollment to hospital discharge or Day 60, whichever is sooner

CONTACTS AND LOCATIONS:
Overall Officials: Hernando Gomez, MD, MPH, Principal Investigator — Center for Critical Care Nephrology, University of Pittsburgh Medical Center
Locations (12):
- United States (3):
  - LSU Health Sciences Center, 1541 Kings Highway, Shreveport, Louisiana
  - Brigham and Womens Hospital, 75 Francis Street, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, New York
- Belgium (2):
  - AZ Sint-Jan Brugge-Oostende, Intensieve Zorgen, Ruddershove 10, Bruges, West-Vlaanderen
  - Hôpital Erasme, Soins Intensifs, Route de Lennik 808, Brussels
- France (4):
  - CHU Angers, 4 Rue Larrey, Angers, Maine-et-Loire
  - Centre Hospitalier de Béthune, Service de Réanimation et Surveillance continue, 27 rue Delbecque, Béthune, Pas-de-Calais
  - CHRU Dijon Complexe Du Bocage, Department Infectiologie, 14 rue Gaffarel, Dijon
  - Hopital Cochin, 27 Rue Du Faubourg Saint Jacques, Paris
- Germany (3):
  - University Clinic Heidelberg, Klinik für Anaesthesiologie, Im Neuenheimer Feld 110, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Leipzig, Klinik und Poliklinik für Anästhesiologie und Intensivtherapie, Liebigstraße 20, Leipzig, Saxony
  - Universitatsklinikum Munster, Albert-Schweitzer-Campus 1, Münster

REFERENCES:
- [Derived] Molinari L, Heskia F, Peerapornratana S, Ronco C, Guzzi L, Toback S, Birch R, Beyhaghi H, Kwan T, Kampf JP, Yealy DM, Kellum JA; Sapphire and Protocolized Care for Early Septic Shock (ProCESS) Investigators. Limiting Acute Kidney Injury Progression In Sepsis: Study Protocol and Trial Simulation. Crit Care Med. 2021 Oct 1;49(10):1706-1716. doi: 10.1097/CCM.0000000000005061. PMID 33927121